CLINICAL TRIAL: NCT01399619
Title: Safety and Efficacy of 120mg and 240mg BI 201335 Once Daily in Combination With Pegylated Interferon Alpha and Ribavirin for Treatment of Chronic Hepatitis C (HCV) Genotype 1 Infection in HIV/HCV Co-infected Patients. A Multinational, Randomised, Parallel Group, Open-label Trial.
Brief Title: Phase III Trial of BI 201335 (Faldaprevir) in Treatment Naive (TN) and Relapser Hepatitis C Virus (HCV)-Human Immunodeficiency Virus (HIV) Coinfected Patients (STARTverso 4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1220.19; 2010-021734-59 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — faldaprevir

ARMS (3):
- BI201335 12W (Experimental): patient to receive two capsules of BI 201335 once a day for 12 weeks and pegIFN/RBV for 24 or 48 weeks
  Interventions: Drug: PegIFN/RBV; Drug: BI201335
- BI 201335 24W (Experimental): patient to receive two capsules of BI 201335 once a day for 24 weeks and PegIFN/RBV for 24 or 48 weeks
  Interventions: Drug: BI201335 24W; Drug: PegIFN/RBV
- BI 201335 24 W (Experimental): patient to receive one capsule of BI 201335 once a day for 24 weeks and pegIFN/RBV for 24 or 48 weeks
  Interventions: Drug: PegIFN/RBV; Drug: Bi 201335

INTERVENTIONS:
Drug: PegIFN/RBV — PegIFN/RBV for 24 or 48w
  Arms: BI 201335 24 W
Drug: PegIFN/RBV — PegIFN/RBV for 24 or 48w
  Arms: BI201335 12W
Drug: BI201335 — BI201335 for 12w
  Arms: BI201335 12W
Drug: BI201335 24W — BI201335 for 24w
  Arms: BI 201335 24W
Drug: PegIFN/RBV — PegIFN/RBV for 24 or 48w
  Arms: BI 201335 24W
Drug: Bi 201335 — BI 201335 for 24 w
  Arms: BI 201335 24 W

SUMMARY:
the aim of this trial is to evaluate the efficacy and the safety of BI 201335 given for 12 or 24 weeks in combination with PegIFN/RBV given for 24-48 weeks, according to re-randomisation of Early Treatment Success (ETS) patients at 24 weeks to stop PegIFN/RBV or continue PegIFN/RBV until week 48. If no ETS, then PegIFN/RB for 48 weeks, in HCV treatment-naive or relapsers patients coinfected with HIV

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C (HCV) genotype 1 infection
2. Chronic Human Immunodeficiency Virus (HIV) -1 infection
3. HCV treatment naive or HCV treatment experienced but only relapsers
4. Age 18 to 70 years
5. Antiretroviral treatment naive or on stable Highly Active Antiretroviral Therapy (HAART)
6. Karnofsky score >70
7. HCV viral load >1.000 IU/mL

Exclusion criteria:

1. HCV infection of mixed genotype (1/2, 1/3, 1/4)
2. Evidence of acute or chronic liver due to chronic HCV infection
3. Hepatitis B virus (HBV) infection with presence of HBs-Ag
4. Active malignancy or history or malignancy within the last 5 years
5. Received concomitant systemic antiviral (other than antiretroviral), hematopoietic growth factor or immunomodulatory treatment in 28 days prior enrolment.
6. Decompensated liver disease,as evidenced by ascites, hepatic encephalopathy, esophageal variceal bleeding, and/or laboratory values that add up to >/= 7 points according tho the Child-Turcotte-Pugh classification
7. Hemoglobin </=11g/dL for women and </= 12 g/dL for men
8. Patients with stable cardiac disease and Hemoglobin <12g/dL
9. Known hypersensitivity to any ingredient of the study drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (71):
- United States (22):
  - 1220.19.0045 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1220.19.0007 Boehringer Ingelheim Investigational Site, Palm Springs, California
  - 1220.19.0031 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1220.19.0005 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1220.19.0086 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1220.19.0044 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1220.19.0004 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 1220.19.0079 Boehringer Ingelheim Investigational Site, Lutherville, Maryland
  - 1220.19.0027 Boehringer Ingelheim Investigational Site, Framingham, Massachusetts
  - 1220.19.0008 Boehringer Ingelheim Investigational Site, Camden, New Jersey
  - 1220.19.0009 Boehringer Ingelheim Investigational Site, Hillsborough, New Jersey
  - 1220.19.0011 Boehringer Ingelheim Investigational Site, Albany, New York
  - 1220.19.0006 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.19.0014 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.19.0084 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.19.0021 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1220.19.0013 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1220.19.0029 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1220.19.0012 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1220.19.0060 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1220.19.0016 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1220.19.0026 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Brazil (6):
  - 1220.19.5508 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 1220.19.5502 Boehringer Ingelheim Investigational Site, Rio de Janeiro - RJ
  - 1220.19.5506 Boehringer Ingelheim Investigational Site, Salvador
  - 1220.19.5503 Boehringer Ingelheim Investigational Site, São Paulo
  - 1220.19.5505 Boehringer Ingelheim Investigational Site, São Paulo
  - 1220.19.5501 Boehringer Ingelheim Investigational Site, São Paulo - SP
- France (6):
  - 1220.19.3306 Boehringer Ingelheim Investigational Site, Lyon
  - 1220.19.3303 Boehringer Ingelheim Investigational Site, Marseille
  - 1220.19.3304 Boehringer Ingelheim Investigational Site, Marseille
  - 1220.19.3301 Boehringer Ingelheim Investigational Site, Paris
  - 1220.19.3305 Boehringer Ingelheim Investigational Site, Paris
  - 1220.19.3307 Boehringer Ingelheim Investigational Site, Paris
- Germany (9):
  - 1220.19.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.19.4921 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.19.4901 Boehringer Ingelheim Investigational Site, Bonn
  - 1220.19.4924 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1220.19.4919 Boehringer Ingelheim Investigational Site, Hamburg
  - 1220.19.4920 Boehringer Ingelheim Investigational Site, Hamburg
  - 1220.19.4905 Boehringer Ingelheim Investigational Site, München
  - 1220.19.4922 Boehringer Ingelheim Investigational Site, München
  - 1220.19.4923 Boehringer Ingelheim Investigational Site, Würzburg
- Italy (7):
  - 1220.19.3901 Boehringer Ingelheim Investigational Site, Antella (fi)
  - 1220.19.3902 Boehringer Ingelheim Investigational Site, Bari
  - 1220.19.3906 Boehringer Ingelheim Investigational Site, Brescia
  - 1220.19.3907 Boehringer Ingelheim Investigational Site, Milan
  - 1220.19.3905 Boehringer Ingelheim Investigational Site, Pavia
  - 1220.19.3903 Boehringer Ingelheim Investigational Site, Roma
  - 1220.19.3904 Boehringer Ingelheim Investigational Site, Torino
- Spain (9):
  - 1220.19.3404 Boehringer Ingelheim Investigational Site, Badalona
  - 1220.19.3401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.19.3403 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.19.3409 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.19.3402 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1220.19.3405 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.19.3406 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.19.3407 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.19.3408 Boehringer Ingelheim Investigational Site, Seville
- Switzerland (4):
  - 1220.19.4101 Boehringer Ingelheim Investigational Site, Basel
  - 1220.19.4103 Boehringer Ingelheim Investigational Site, Bern
  - 1220.19.4102 Boehringer Ingelheim Investigational Site, Lugano
  - 1220.19.4104 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (8):
  - 1220.19.4406 Boehringer Ingelheim Investigational Site, Brighton
  - 1220.19.4407 Boehringer Ingelheim Investigational Site, Edinburgh
  - 1220.19.4401 Boehringer Ingelheim Investigational Site, London
  - 1220.19.4402 Boehringer Ingelheim Investigational Site, London
  - 1220.19.4403 Boehringer Ingelheim Investigational Site, London
  - 1220.19.4404 Boehringer Ingelheim Investigational Site, London
  - 1220.19.4408 Boehringer Ingelheim Investigational Site, London
  - 1220.19.4405 Boehringer Ingelheim Investigational Site, Manchester

REFERENCES:
- [Derived] Dieterich D, Nelson M, Soriano V, Arasteh K, Guardiola JM, Rockstroh JK, Bhagani S, Laguno M, Tural C, Ingiliz P, Jain MK, Stern JO, Manero M, Vinisko R, Kort J; STARTVerso4 study group. Faldaprevir and pegylated interferon alpha-2a/ribavirin in individuals co-infected with hepatitis C virus genotype-1 and HIV. AIDS. 2015 Mar 13;29(5):571-81. doi: 10.1097/QAD.0000000000000579. PMID 25710287

RESULTS

PARTICIPANT FLOW:
Groups:
- Faldaprevir 120mg -24W: Faldaprevir (BI 201335) 120 mg once a day (QD) combined with pegIFN/RBV for 24 weeks, at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
- Faldaprevir 240mg -12W: Faldaprevir 240 mg QD plus pegIFN/RBV for 12 weeks followed by re-randomisation at Week 12 to stop Faldaprevir and continue pegIFN/RBV alone until Week 24; at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
- Faldaprevir 240mg-24W: Faldaprevir 240 mg QD plus pegIFN/RBV for 12 weeks followed by re-randomisation at Week 12 to continue Faldaprevir to Week 24, at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
- Faldaprevir 240 mg -NR (Prior to Re-randomization at Week 12): Patients initially assigned to Faldaprevir 240 mg who discontinued prior to re-randomization at WK 12.
Period: Overall Study
Arm/Group | Faldaprevir 120mg -24W | Faldaprevir 240mg -12W | Faldaprevir 240mg-24W | Faldaprevir 240 mg -NR (Prior to Re-randomization at Week 12)
Started | 123 | 84 | 86 | 17
Completed | 98 | 84 | 74 | 0
Not Completed | 25 | 0 | 12 | 17
Not completed — Adverse Event | 10 | 0 | 4 | 10
Not completed — Lack of Efficacy | 9 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 3 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Not treated | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: FAS (All patients who were randomized and received at least one dose of assigned therapy)
Groups:
- Faldaprevir 120mg - 24W: Faldaprevir 120 mg QD combined with pegIFN/RBV for 24 weeks, at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
- Faldaprevir 240mg -T: patient to receive Faldaprevir 240 mg once a day for 12 or 24 weeks and PegIFN/RBV for 24 or 48 weeks + patients who received Faldaprevir 240 mg and discontinued prior to week 12.
- Total: Total of all reporting groups
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg -T | Total
Number analyzed (Participants) | 123 | 185 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (7.63) | 46.5 (8.36) | 46.9 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 40 | 60
  Male | 103 | 145 | 248

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR12)
Description: Percentage of participants with sustained Virological Response SVR12: Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) level <25 IU/mL, undetected 12 weeks after the planned end of treatment.
Time Frame: 60 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Faldaprevir 120mg - 24W: Faldaprevir 120 mg once a day (QD) combined with pegIFN/RBV for 24 weeks, at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
- Faldaprevir 240mg - 12W: Faldaprevir 240 mg QD plus pegIFN/RBV for 12 weeks followed by re-randomisation at Week 12 to stop Faldaprevir and continue pegIFN/RBV alone until Week 24; at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
- Faldaprevir 240mg - 24W: Faldaprevir 240 mg QD plus pegIFN/RBV for 12 weeks followed by re-randomisation at Week 12 to continue BI 201335 to Week 24, at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
- Faldaprevir 240mg -T: Faldaprevir 240mg-12w + Faldaprevir 240mg-24w + patients initially randomized or assigned to Faldaprevir 240 mg who discontinued prior to re-randomization at Week 12.
- Faldaprevir - Total: Total subjects who were treated with Faldaprevir.
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
percentage of participants | 70.7 [62.7 to 78.8] | 78.6 [69.8 to 87.3] | 76.7 [67.8 to 85.7] | 72.4 [66.0 to 78.9] | 71.8 [66.7 to 76.8]
Statistical Analysis 1: Comparison: Faldaprevir - Total; the SVR12 rate in total Faldaprevir group compared with the historical rate of 40%; Test type: Superiority or Other; p < 0.0001, normal approximation — p-value corresponds to a two sided test against the historical rate of 40%

2. Secondary Outcome: Virological Response 24 Weeks Post Treatment (SVR24)
Description: Percentage of participants with virological response 24 weeks post treatment (SVR24): Plasma HCV RNA level<25IU/mL (undetected) 24 weeks after the planned end of treatment.
Time Frame: 72 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Faldaprevir 240mg - 24W: Faldaprevir 240 mg QD plus pegIFN/RBV for 12 weeks followed by re-randomisation at Week 12 to continue Faldaprevir to Week 24, at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
percentage of participants | 69.9 [61.8 to 78.0] | 78.6 [69.8 to 87.3] | 74.4 [65.2 to 83.6] | 71.4 [64.8 to 77.9] | 70.8 [65.7 to 75.9]

3. Secondary Outcome: Early Treatment Success (ETS)
Description: Early Treatment Success (ETS): Plasma HCV RNA level<25 IU/mL (detected or undetected) at Week 4 and HCV RNA< 25 IU/mL, undetected at Week 8
Time Frame: Week 4, week 8 and week 60
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg -12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  number of subjects with ETS =yes | 95 | 70 | 73 | 150 | 245
  number of subjects with SVR12 among ETS=yes group | 83 | 62 | 63 | 127 | 210

4. Secondary Outcome: The Number of Participants With Alanine Aminotransferase (ALT) Normalisation at End of Treatment (EoT) When SVR12=Yes
Description: The number of participants with Alanine Aminotransferase (ALT) normalisation at End of Treatment (EoT) when SVR12=yes. BL stands for baseline.
Time Frame: 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=yes | 87 | 66 | 66 | 134 | 221
  SVR12=yes, BL normal to EOT normal | 29 | 16 | 26 | 43 | 72
  SVR12=yes, BL elevated to EOT normal | 45 | 34 | 32 | 66 | 111
  SVR12=yes, No BL or EoT data | 0 | 0 | 0 | 1 | 1

5. Secondary Outcome: The Number of Participants With Alanine Aminotransferase (ALT) Normalisation at End of Treatment When SVR12=no
Description: The number of participants with Alanine Aminotransferase (ALT) normalisation: ALT in normal range at End of Treatment when SVR12=no. BL stands for baseline.
Time Frame: 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg -12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=no | 36 | 18 | 20 | 51 | 87
  SVR12=no, BL normal to EoT normal | 18 | 5 | 5 | 18 | 36
  SVR12=no, BL elevated to EoT normal | 12 | 8 | 9 | 21 | 33
  SVR12=no, no BL or EoT data available | 2 | 0 | 0 | 0 | 2

6. Secondary Outcome: The Number of Participants With Alanine Aminotransferase (ALT) Normalisation at Post Treatment When SVR12=Yes
Description: The number of participants with ALT in normal range at post treatment (SVR12 Visit) when SVR12=yes. BL = baseline.
Time Frame: 60 weeks
Population: FAS
Measure: Number; unit: participants
Groups:
- Faldaprevir 120mg -24W: Faldaprevir 120 mg once a day (QD) combined with pegIFN/RBV for 24 weeks, at Week 24, randomisation of patients who achieved early treatment success (ETS) to an additional 24 weeks of pegIFN/RBV or to stop treatment; patients who did not achieve ETS received pegIFN/RBV until Week 48.
Arm/Group | Faldaprevir 120mg -24W | Faldaprevir 240mg -12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=yes | 87 | 66 | 66 | 134 | 221
  SVR12=yes, BL normal to SVR12 normal | 28 | 17 | 26 | 45 | 73
  SVR12=yes, BL elevated to SVR12 normal | 52 | 46 | 35 | 81 | 133
  SVR12=yes, no ALT data available at SVR12 visit | 4 | 0 | 1 | 1 | 5

7. Secondary Outcome: The Number of Participants With Alanine Aminotransferase (ALT) Normalisation at Post Treatment When SVR12=no
Description: The number of participants with ALT in normal range at post treatment (SVR12 Visit) when SVR12=no. BL = baseline.
Time Frame: 60 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=no | 36 | 18 | 20 | 51 | 87
  SVR12=no, BL normal to SVR12 normal | 8 | 1 | 3 | 6 | 14
  SVR12=no, BL elevated to SVR12 normal | 1 | 6 | 3 | 9 | 10
  SVR12=no, no ALT data available at SVR12 visit | 16 | 4 | 6 | 20 | 36

8. Secondary Outcome: The Number of Participants With Aspartate Aminotransferase (AST) Normalisation at End of Treatment When SVR12=Yes
Description: The number of participants with Aspartate Aminotransferase (AST) normalisation at End of Treatment when SVR12=yes. BL = baseline.
Time Frame: 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=yes | 87 | 66 | 66 | 134 | 221
  SVR12=yes, BL normal to EoT normal | 41 | 25 | 28 | 54 | 95
  SVR12=yes, BL elevated to EoT normal | 32 | 25 | 27 | 52 | 84
  SVR12=yes, no BL or EoT data available | 0 | 0 | 0 | 1 | 1

9. Secondary Outcome: The Number of Participants With Aspartate Aminotransferase (AST) Normalisation at End of Treatment When SVR12=no
Description: The number of participants with Aspartate Aminotransferase (AST) normalisation at End of Treatment when SVR12=no. BL = baseline.
Time Frame: 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=no | 36 | 18 | 20 | 51 | 87
  SVR12=no, BL normal to EoT normal | 14 | 6 | 7 | 19 | 33
  SVR12=no, BL elevated to EoT normal | 12 | 6 | 8 | 19 | 31
  SVR12=no, no BL or EoT data available | 2 | 0 | 0 | 0 | 2

10. Secondary Outcome: The Number of Participants With Aspartate Aminotransferase (AST) Normalisation at Post Treatment When SVR12=Yes
Description: The number of participants with AST in normal range at Post Treatment (SVR12 Visit) when SVR12=yes. BL = baseline.
Time Frame: 60 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=yes | 87 | 66 | 66 | 134 | 221
  SVR12=yes, BL normal to SVR12 normal | 41 | 27 | 28 | 57 | 98
  SVR12=yes, BL elevated to SVR12 normal | 36 | 36 | 33 | 69 | 105
  SVR12=yes, no AST data available at SVR12 visit | 4 | 0 | 1 | 1 | 5

11. Secondary Outcome: The Number of Participants With Aspartate Aminotransferase (AST) Normalisation at Post Treatment When SVR12=no
Description: The number of participants with AST in normal range at Post Treatment (SVR12 Visit) when SVR12=no. BL = baseline.
Time Frame: 60 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T | Faldaprevir - Total
Number analyzed (Participants) | 123 | 84 | 86 | 185 | 308
participants
  SVR12=no | 36 | 18 | 20 | 51 | 87
  SVR12=no, BL normal to SVR12 normal | 6 | 4 | 6 | 13 | 19
  SVR12=no, BL elevated to SVR12 normal | 2 | 3 | 0 | 3 | 5
  SVR12=no, no AST data available at SVR12 visit | 16 | 4 | 6 | 20 | 36

ADVERSE EVENTS:
Time Frame: from the start date of trial medication up to 52 weeks ( AEs occurred from the start date of trial medication up to four weeks after all treatment discontinuation).
Arm/Group | Faldaprevir 120mg - 24W | Faldaprevir 240mg - 12W | Faldaprevir 240mg - 24W | Faldaprevir 240mg -T
Serious Adverse Events (participants affected / at risk) | 17/123 | 5/84 | 5/86 | 15/185
Other Adverse Events (participants affected / at risk) | 116/123 | 80/84 | 84/86 | 178/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120mg - 24W (N=123) | Faldaprevir 240mg - 12W (N=84) | Faldaprevir 240mg - 24W (N=86) | Faldaprevir 240mg -T (N=185)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0 | 0 | 0
Leishmaniasis (Infections and infestations) | 0 | 0 | 1 | 1
Neurosyphilis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Substance use (Social circumstances) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120mg - 24W (N=123) | Faldaprevir 240mg - 12W (N=84) | Faldaprevir 240mg - 24W (N=86) | Faldaprevir 240mg -T (N=185)
Anaemia (Blood and lymphatic system disorders) | 27 | 13 | 15 | 30
Neutropenia (Blood and lymphatic system disorders) | 27 | 6 | 15 | 22
Dry eye (Eye disorders) | 3 | 5 | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 7 | 11 | 4 | 17
Abdominal pain upper (Gastrointestinal disorders) | 7 | 7 | 3 | 10
Cheilitis (Gastrointestinal disorders) | 8 | 4 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 31 | 24 | 23 | 51
Dry mouth (Gastrointestinal disorders) | 6 | 5 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 6 | 4 | 7 | 11
Nausea (Gastrointestinal disorders) | 34 | 38 | 36 | 81
Vomiting (Gastrointestinal disorders) | 12 | 14 | 23 | 43
Asthenia (General disorders) | 31 | 21 | 17 | 39
Chills (General disorders) | 5 | 2 | 7 | 11
Fatigue (General disorders) | 39 | 29 | 30 | 65
Influenza like illness (General disorders) | 14 | 17 | 12 | 31
Injection site reaction (General disorders) | 3 | 2 | 6 | 8
Irritability (General disorders) | 19 | 8 | 5 | 13
Pyrexia (General disorders) | 29 | 11 | 10 | 24
Jaundice (Hepatobiliary disorders) | 7 | 8 | 10 | 19
Oral herpes (Infections and infestations) | 8 | 0 | 2 | 2
Weight decreased (Investigations) | 16 | 10 | 13 | 25
Decreased appetite (Metabolism and nutrition disorders) | 29 | 14 | 18 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6 | 6 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 9 | 15 | 27
Dizziness (Nervous system disorders) | 9 | 10 | 6 | 20
Headache (Nervous system disorders) | 29 | 21 | 22 | 47
Lethargy (Nervous system disorders) | 1 | 3 | 5 | 8
Anxiety (Psychiatric disorders) | 9 | 5 | 2 | 8
Depressed mood (Psychiatric disorders) | 6 | 4 | 7 | 12
Depression (Psychiatric disorders) | 11 | 9 | 13 | 24
Insomnia (Psychiatric disorders) | 29 | 11 | 14 | 28
Sleep disorder (Psychiatric disorders) | 4 | 3 | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 10 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 8 | 3 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 4 | 6 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 9 | 18 | 27
Erythema (Skin and subcutaneous tissue disorders) | 8 | 5 | 5 | 10
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 6 | 3 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 16 | 17 | 34
Rash (Skin and subcutaneous tissue disorders) | 22 | 16 | 13 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.